CLINICAL TRIAL: NCT01074775
Title: An Investigation Of In Vivo Human Innate Immune Responses To Mycobacterial Aerodigestive Tract Infection
Brief Title: Human Innate Immune Responses To Mycobacterial Aerodigestive Tract Infection
Acronym: UBC-INNATE01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: University of British Columbia (Other); Wellcome Trust (Other); Fundação Ataulpho de Paiva, Rio de Janeiro, Brasil (Unknown); Foundation for the National Institutes of Health (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: David JM Lewis, St George's, University of London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UBC-INNATE01
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Bacterial Infections
Keywords: innate immunity; mycobacterium bovis; mucosal immunity; adaptive immunity; genomics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Challenge group (Experimental): Recipients of three challenge infections with oral M bovis
  Interventions: Biological: Gut infection challenge with M bovis

INTERVENTIONS:
Biological: Gut infection challenge with M bovis — Oral delivery of 100mg viable M bovis (approximately 10,000,000 viable bacilli) in 5mL 1.5% sodium glutamate solution on three occasions on days 0, 28 and 49
  Other Names: Bacille Calmette Guerin "Moreau Rio de Janeiro"

SUMMARY:
The approach we will use is to employ measurement of the activation of white blood cells, to look at patterns of responses during a controlled infection of the gut with Mycobacterium bovis. M. bovis can be conveniently obtained in a safe and pure form as an oral vaccine. By giving three challenges of M bovis to the gut, we will simulate repeated gut infections with this organism. We can then compare the activation of cells in the blood to the immune responses seen after each challenge, to determine whether the non-specific defences of the gut can block each subsequent infection.

DETAILED DESCRIPTION:
The approach we will use is to employ immune readouts and genomics to look at patterns of responses during a controlled infectious challenge of the human gut.

Genomics uses 'Affymetrix' gene arrays, and other techniques to determine the profile of gene expression. When a gene is 'switched on' it makes mRNA that the body uses as a template to make proteins. We will extract all the mRNA from white blood cells before, during and after an infection. The gene chips have hundreds or thousands of mini-sensors that can measure how much mRNA from any particular gene is present in the sample. Thus we can begin to see which genes are switch on or off, or unaffected, inside white blood cells during the stages of a developing innate immune response. This allows us to monitor the body's response to an infection and to see which families of genes are important at the different stages of gut infection.

The BCG vaccine is derived from Mycobacterium bovis (the full name of the organism is Mycobacterium bovis Baccille Calmette Guérin). In this study we propose to use an oral BCG preparation, produced as a prophylactic and therapeutic oral vaccine, as a safe model for natural gut infection with pathogenic Mycobacterium bovis. The cell wall of mycobacteria such as BCG is a powerful immune adjuvant (an adjuvant is a substance that enhances an immune response) as the lipids, sugars and proteins in the cell wall interact strongly with the molecules of the innate immune system. It therefore provides a safe but highly effective way to stimulate innate immunity under 'natural' conditions of gut infection. This first model has been selected as it reflects a 'real world' high priority area of disease prevention, while having a high level of safety and reproducibility in the oral BCG model.

By carefully delivering oral BCG challenges to healthy volunteers under controlled conditions, we can reduce the noise and background activity in the proteomic and genomic assays we will use to profile the developing innate immune response. We can check that the BCG has indeed colonised and 'infected' the subject by measuring the specific adaptive T cell and antibody responses using sensitive assays we have developed in previous studies to detect these immune responses. This is a critical aspect of the study: if we detect the BCG-specific T cell responses we can be assured that the 'infection' has taken place, and so can interpret the profiles we see in the immunology and genomics.

If we see an immune response we can relate any innate immune activation to colonisation with BCG. In contrast, even if we see no immune responses, but can be sure that the vaccine was delivered properly in a viable formulation (which we will do by adhering to strict Good Clinical Practice) then we can look at features in the genomic and proteomic profiles in the baseline measurements before infection that may predict the failure of the organisms to infect.

By collecting data of other events such as intercurrent illnesses, or other adverse events we can also determine whether changes in the proteomic or gene expression profiles are indeed due to the model infection, or extraneous events. This preliminary study will enable us to refine expensive techniques, protocols and assays to let us focus in more detail in subsequent studies

This study will be conducted according to the Standard Operating Procedures (SOPs) of the St George's Vaccine Institute. Up to 10 subjects will be included in this study. The study will consist of a pre-study screening visit and 23 visits over a period of 12 month at the times indicated in the schedule for investigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers, 18 to 45 years of age, who sign an informed consent form following a detailed explanation of participation in the protocol.
* Volunteers who are in good health as determined by medical history, physical examination and clinical judgement.
* Volunteers who will be available for the duration of the study.
* Volunteers willing and able to give written informed consent.

Exclusion Criteria:

* Volunteers who are contraindicated for BCG vaccination according to the Manufacturer's Data Sheet.
* Individuals who have hypersensitivity to any component of the vaccine used in this study.
* Individuals who have severe or multiple allergies, including to drugs or pharmaceutical agents.
* Volunteers who are receiving drug treatment for, or who have a significant history of, cardiological or respiratory disease. Volunteers who are suffering from severe cardio-respiratory disease, including hypertension, or an active neurological disorder.
* Individuals found to be HIV antibody positive at screening, or with a known impairment of immune function, or those receiving immunosuppressive therapy, including regular inhaled steroids. Intermittent steroid use (less than twice per month in the preceding 3 months) is acceptable.
* Individuals with acute infections (including fever >38°C).
* Women who are pregnant or lactating.
* Women capable of becoming pregnant who do not agree to have pregnancy testing before immunisation, and/or who do not agree to take effective contraception for the duration of the study period.
* Individuals with a current problem with substance abuse or with a history of substance abuse, which, in the opinion of the investigator, might interfere with participation in the study.
* Individuals with any condition, which, in the opinion of the investigator, might interfere with the evaluation with the study objectives.
* Individuals who have received an investigational agent within 30 days prior to entry, or been in any other study in the last 6 months.
* Individuals who are planning to leave the area of the study site prior to the end of the study period, or who are likely not to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Genomics profile | 12 months (23 visits)
  Peripheral blood mononuclear cell gene expression measured by analysis of extracted mRNA using polymerase chain reaction

SECONDARY OUTCOMES:
Cell mediated immune responses | 12 months (8 visits)
  Frequency of mycobacterium antigen-specific Interferon gamma producing cells measured in vitro by ELISpot and ELISA

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's - University of London, UK
Locations (1):
- St George's Vaccine Institute, St George's University of London, London, England, United Kingdom

REFERENCES:
- See also: St George's Vaccine Institute website — http://www.vaccine.ac.uk
- See also: St George's - University of London website — http://www.sgul.ac.uk